CLINICAL TRIAL: NCT04783298
Title: Can Methods From Computational Psychology be Used to Phenotype Individuals Most Likely to be Non-adherent to Fitness Goals?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dublin City University (Other)
Responsible Party: Sponsor
Other Study IDs: DCUSOC29012021MMCC1
Record Dates: First submitted 2021-02-15; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Lifestyle, Sedentary
MeSH Terms: conditions — Sedentary Behavior | interventions — Amyloid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: App — An application to deliver a series of behavioral questionnaires and decision-making game

SUMMARY:
This is a longitudinal study combining objective sensor data, with decision-making games and contextual personality traits to identify patterns in exercise decay. The data generated will be used to build computational models to predict digital personas, and help identify those individuals most likely to abandon exercise goals.

DETAILED DESCRIPTION:
Interested individuals to be recruited on social media and invited to download the study app. The plain language statement and informed consent are embedded in the app. Once e-consent is obtained, individuals will share their Fitbit data and complete the following questionnaires; Type D Personality, Goal Setting, and Self-Efficacy questionnaire and a decision-making game based on the IGT. After a 6 month time period, they will be requested to retake the questionnaires and decision-making game.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals who have a Fitbit

Exclusion Criteria:

* Individuals under the age of 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals starting a new exercise regime.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity measured by an increase in weekly steps measured by Fitbit. | Week 1 and 6 months
  Fitbit is a physical activity tracker worn on the wrist and objectively measures steps taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Dublin City University, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCarthy M, Zhang L, Monacelli G, Ward T. Using Methods From Computational Decision-making to Predict Nonadherence to Fitness Goals: Protocol for an Observational Study. JMIR Res Protoc. 2021 Nov 26;10(11):e29758. doi: 10.2196/29758. PMID 34842557